CLINICAL TRIAL: NCT03169322
Title: Influence of Mouth Breathing on Outcome of Scaling and Root Planing in Chronic Periodontitis
Brief Title: Influence of Mouth Breathing on Periodontal Healing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Manpreet Perio
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Active Comparator): patients having chronic periodontitis with mouth breathing habit will receive scaling and root planing (SRP)
  Interventions: Procedure: SRP
- Control Group (Active Comparator): Nose breathers having chronic periodontitis will receive scaling and root planing (SRP)
  Interventions: Procedure: SRP

INTERVENTIONS:
Procedure: SRP — patients having chronic periodontitis with mouth breathing habit will receive scaling and root planing

SUMMARY:
Studies reveal association between dry conditions and decreased healing in wounds or any treatment. From these studies, it can be hypothesized that healing in mouth breathers after scaling and root planing in terms of bleeding on probing, gingival index, plaque Index, clinical attachment level, probing depth may not show as much improvement as in case of nose breathers. No study has been conducted till date to find effect of scaling and root planing in periodontitis patients among mouth breathers and nose breathers.

DETAILED DESCRIPTION:
INTRODUCTION

Mouth breathing is perceived to be responsible for persistant marginal gingivitis. The most common region to be affected by gingivitis in mouth breathers is maxillary anterior region. Other areas are affected in following decreasing order: maxillary posterior areas, mandibular anterior region and mandibular posterior region. Various reasons are considered to be responsible for gingival inflammation in mouth breathers. Possible factors responsible for gingival inflammation may be continuous loss of saliva over marginal tissues leading to increased plaque scores or qualitative change in plaque in terms of incorporation of more virulent strains of bacteria in plaque.

Mouth breathing, lip seal, upper lip coverage are related. In one study, mouth breathing along with incompetent lip seal and decreased upper lip coverage were associated with gingivitis. In other study plaque was thought to be a contributing factor for gingivitis in patients with decreased upper lip coverage. One study showed lack of lip seal due to increased overjet to be responsible for increased gingival inflammation. Kolawole KA et al in their study found that lip incompetence was associated with increased plaque scores. It may be due to lack of normal cleansing action of saliva. No association between mouth breathing and gingivitis prevalence had been reported in the study by Sutcliffe. However mouth breathing slightly increased severity of gingivitis.

Saliva performs very important functions including lubrication of oral tissues, antimicrobial action, regulation of pH, elimination of food bolus and facilitating in removal of carbon. Salivary flow provides mechanical cleansing of residues present in mouth such as non adherent bacteria, cellular and food debris. Lack of salivary flushing action results in accumulation of food debris and dental plaque thus promoting an acidogenic and aciduric oral bacteria responsible for dental caries.

Xerostomia /dry mouth is responsible for increase in gingival inflammation and also affects periodontal conditions with increased probing depth, plaque index. In one study, young adults with self reporting of xerostomia had increased sites with bleeding on probing and increased plaque scores. Proliferative activity of oral gingival epithelium is decreased in inflamed gingiva of patients with xerostomia. In one study, healing in gingivectomy wound was delayed in sialadenectomized rats.

In habitual mouth-breathers, 50% of the inspired air passes through mouth. In mouth-breathers, amount of water evaporated from saliva into air may reach 0.24 mL/min resulting in greater retention of bacteria in oral cavity.

For transient relief of xerostomia, salivary substitutes and sugar free gums and lozenges are available. Effect of salivary substitutes along with scaling and root planing in mouth breathers have been evaluated in one study. It was found that in mouth breathers, scaling and root planing along with application of salivary substitutes provided better improvement in gingival index, bleeding on probing, clinical attachment level than in whom scaling and root planing alone was performed.

Better response of gingiva was seen in mouth breathers after 4-6 weeks of oral debridement and use of petroleum jelly. However when use of petroleum jelly was withheld inflammation was again noticed in gingiva.

Similar effects of drying conditions are seen in various parts of body. In children with dry skin and predisposition to atopic dermatitis, use of emollients was seen to improve their skin conditions.

All these studies reveal association between dry conditions and decreased healing in wounds or any treatment. From these studies, it can be hypothesized that healing in mouth breathers after scaling and root planing in terms of bleeding on probing, gingival index, plaque Index, clinical attachment level, probing depth may not show as much improvement as in case of nose breathers. No study has been conducted till date to find effect of scaling and root planing in periodontitis patients among mouth breathers and nose breathers.

MATERIAL AND METHODS

This study will be conducted in Department of Periodontics, Post Graduate Institute of Dental Sciences(PGIDS), Rohtak.

STUDY POPULATION AND DESIGN

Patients suffering from chronic periodontitis of age group 20-35 years will be recruited from regular OPD of the Department of Periodontics in the study. Approximately 60 patients would comprise test group and control group. Test group (n≈30) will include individuals having mouth breathing habit. Control group (n≈30) will comprise of patients who are nose breathers.

METHODOLOGY

The study will be conducted in accordance with the ethical standards outlined in the 1964 Declaration of Helsinki, as revised in 2013.

Diagnosis of mouth breathing

Diagnosis of mouth breathing will be made on the basis of patient history. Patients would be asked whether, in their opinion, they are mouth breathers, and also whether they have dry mouth on awakening.

Study groups

After carefully explaining the nature and objectives of the study, written informed consent will be obtained from each patient of study group.

Participants belonging to both study groups would receive conventional periodontal treatment, i.e. scaling and root planing (SRP).

Clinical measurement

All of the participants will undergo full mouth examination in a standardized way using illumination by a standard dental light, a mouth mirror, explorer and University of North Carolina -15(UNC-15) periodontal probe and the following parameters will be recorded: plaque index (PI), gingival index (GI), bleeding on probing (BOP), probing depth (PD), and clinical attachment level (CAL). Degree of maxillary incisor coverage by upper lip at rest would be classified into 2 types: total coverage, maxillary labial gingiva exposed. Teeth will be assessed at four sites for PI and GI, and at six sites for PD, CAL, and BOP during full mouth periodontal examination. BOP will be assessed as a dichotomous measure within 15 seconds of probing to full pocket depth. After the initial readings for PI, GI, BOP, PD, CAL at baseline will be recorded; patients would receive oral hygiene instructions and full-mouth SRP. Patients will be re-examined at 4th, 8th, 12th week. Reinforcement of oral hygiene will be carried out at each recall visit. PI, BOP and GI will be recorded at 4, 8 and 12 weeks of treatment. The other parameters would be measured only at the completion of 12 weeks of SRP.

All clinical periodontal examinations will be carried out by a single investigator to preclude any inter-examiner variability.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy individuals possessing ≥ 20 natural teeth.
* Chronic periodontitis criteria as defined by division of Oral Health at the Centre for Disease Control and Prevention(CDC) in collaboration with American Academy of Periodontology(AAP)-(Page and Eke 2012) i.e. at least two or more interproximal sites with clinical attachment loss(CAL) ≥ 4mm(not on same tooth), or ≥2 interproximal sites with Pocket Depth(PD) ≥5 mm(not on same tooth).
* BOP prevalence >25%.

Exclusion Criteria:

* Patients on anti-inflammatory drugs or antibiotics within previous 6 months of commencement of study, or on any other regular medication or mouth wash, that is likely to influence periodontal status.
* History of periodontal treatment within 1 year of inclusion in the study.
* Current or former smokers or use of tobacco in any form.
* History of treatment with statins, glucocorticoids, anticoagulants, phenytoin, calcium channel blockers such as nifedipine, diltiazem, verapamil, felodipine; immunosuppressants such as cyclosporine; bisphosphonates or any other host modulatory drugs during last six months.
* Non-plaque-induced gingival lesions.
* Patients taking drugs reported to cause xerostomia such as anti-cholinergics, anti-hypertensives, analgesics, sedatives, tranquilizing agents, antihistamines.
* A recent history of any other acute or chronic infection.
* Pregnant and lactating women and those taking oral contraceptive drugs.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-10-14 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
BOP (Bleeding on probing) | 12 Weeks
  Bleeding on probing Bleeding on probing (BOP) has been used to clinically characterize the degree of gingival /periodontal inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Manpreet Kaur, Principal Investigator — Post Graduate Institute of Dental Sciences, Rohtak. HARYANA .INDIA
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: Yes